CLINICAL TRIAL: NCT04066777
Title: The Effect of Alcohol Septal Ablation Therapy on Left Ventricular Function and Invasive Hemodynamics at Rest and During Exercise in Patients With Hypertrophic Obstructive Cardiomyopathy
Brief Title: The Effect of TASH in Patients With HOCM
Acronym: Post-TASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steen Hvitfeldt Poulsen (Other)
Responsible Party: Sponsor-Investigator, Steen Hvitfeldt Poulsen, professor, Aarhus University Hospital Skejby
Organization: Aarhus University Hospital Skejby (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-62-19
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Hypertrophic Obstructive Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic | interventions — Ethanol

STUDY DESIGN:
Intervention Model Description: prospective controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypertrophic obstructive cardiomyopathy (Other): injection of 1-4 mL of 96% ethanol into a septal perforator of the left anterior coronary artery to produce a myocardial infarction
  Interventions: Procedure: alcohol septal ablation

INTERVENTIONS:
Procedure: alcohol septal ablation — injection of 1-4 mL of 96% ethanol into a septal perforator of the left anterior coronary artery to produce a myocardial infarction

SUMMARY:
To examine patients with hypertrophic obstructive cardiomyopathy (HOCM) before and after septal alcohol ablation, to investigate the effect of the treatment in regards to changes in myocardial function, perfusion, invasive hemodynamics and exercise tolerance.

DETAILED DESCRIPTION:
Patients with HOCM who develop symptoms of heart failure are treated initially with non-vasodilating ß-blockers or verapamil to decrease myocardial contractility and heart rate. A substantial part of patients remain symptomatic despite medical treatment. In these patients interventional or surgical treatments (septal reduction therapies (SRT)) to reduce left ventricular outflow tract obstruction (LVOTO) is considered in the presence of moderate to-severe symptoms (New York Heart Association - functional class (NYHA) III-IV) and/or recurrent exertional syncope and an LVOTO gradient ≥50 mm Hg. In some centers, invasive therapy is also considered in patients with mild symptoms (NYHA Class II) who have a resting or maximum provoked gradient of ≥50 mm Hg (with exercise or Valsalva's maneuver) and moderate-to-severe mitral valve regurgitation. Advanced treatment options are alcohol septal ablation (ASA) or surgical myectomy often combined with mitral valve reconstructive surgery. These treatments have similar outcomes in terms of gradient reduction, symptom improvement and exercise capacity

No previous trials have examined the effect of ASA in HOCM with respect to changes in central hemodynamics and myocardial performance during exercise.

24 HOCM patients will be examined prior to ASA, and approximately six-nine months after ASA.

The examination set-up consists of simultaneous 1) transthoracic echocardiography (TTE), 2) right heart catheterization (RHC) and 3) cardiopulmonary exercise test (CPX).

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular wall thickness ≥ 15 mm in one or more myocardial segments that is not explained by loading conditions
* LVOT gradients ≥ 30 mmHg at rest and/or ≥ 50 mmHg at Valsalva's maneuver or exercise
* NYHA ≥ III

Exclusion Criteria:

* < 18 years
* Fertile women who do not use anti-contraceptives
* Pregnancy
* Patients are allowed to have a pacemaker (eg. an implantable cardioverter defibrillator (ICD)) but cannot be pace-dependent
* Amiodarone treatment
* Persistent or permanent atrial fibrillation/flutter
* Previous SRT
* Alcohol or drug abuse
* Significant co-morbidity (judged by the investigator)
* Patients who cannot give valid consent (e.g. mental illness or dementia) or who do not understand Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Pulmonary capillary wedge pressure (PCWP) during exercise | Changes will be evaluated after an expected average of 6-9 months after treatment
  Change in PCWP at 75 watt (or maximum exercise, if this is < 75 W)

SECONDARY OUTCOMES:
Pulmonary capillary wedge pressure (PCWP) at rest | Changes will be evaluated after an expected average of 6-9 months after treatment
  Changes in PCWP at rest
Peak oxygen uptake (VO2-max) | Changes will be evaluated after an expected average of 6-9 months after treatment
  Changes in maximal oxygen consumption (L/min) measured during cardiopulmonary exercise test
Work capacity | Changes will be evaluated after an expected average of 6-9 months after treatment
  work capacity measured in watt during a cardiopulmonary exercise test
LVOT gradient during maximum exercise | Changes will be evaluated after an expected average of 6-9 months after treatment
  Changes of the LVOT gradient during maximum exercise, measured in mmHg during 2D echocardiography
Coronary flow reserve | Changes will be evaluated after an expected average of 6-9 months after treatment
  Changes in the ratio of maximum coronary blood flow (induced by infusion of adenosin) to resting coronary blood flow, estimated by 2D doppler echocardiography
Changes in biomarkers | Changes will be evaluated after an expected average of 6-9 months after treatment
  Changes in N-terminal pro-brain natriuretic peptide (NT-proBNP) ng/l and troponin T ng/l
Change in GLS (%) at peak exercise | Changes will be evaluated after an expected average of 6-9 months after treatment
  Change in global longitudinal strain (GLS) in % at peak exercise
Changes of symptoms and quality of life estimated by KCCQ | Changes will be evaluated after an expected average of 6-9 months after treatment
  Changes of symptoms and quality of life with Kansas City Cardiomyopathy Questionnaire (KCCQ) assessed by clinical evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Steen Hvitfeldt Poulsen, DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Cardiology, Aarhus N, Danmark, Denmark